CLINICAL TRIAL: NCT06118138
Title: Observational Study of Hyperbaric High Pressure Oxygen Therapy (HBOT) in Patients with Post-COVID Syndrome (PCS) and Myalgic Encephalomyelitis/chronic Fatigue Syndrome (ME/CFS)
Brief Title: Hyperbaric High Pressure Oxygen Therapy in Post-COVID Syndrome and ME/CFS
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: KLINIK BAVARIA Kreischa (Unknown); Vivantes Klinikum im Friedrichshain (Unknown)
Responsible Party: Principal Investigator, Carmen Scheibenbogen, Director of the Institute for Medical Immunology, Charite University, Berlin, Germany
Other Study IDs: HBOT; 01EP2201 (Other Grant/Funding Number: BMBF)
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-09

CONDITIONS: Post-COVID ME/CFS
Keywords: Post-COVID Syndrome; Long COVID; Chronic Fatigue Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Combination Product: Hyperbaric oxygen therapy (HBOT) — HBOT is a medical treatment employed for various conditions. It entails breathing 100% oxygen within a pressurized chamber known as a hyperbaric chamber. This oxygen-rich environment promotes healing and aids in combating specific infections.
  In this study, the investigators will administer HBOT using a hyperbaric chamber set to 2 times the normal atmospheric pressure, indicated as 2 atmosphere absolute (ATA). This pressure surge enhances oxygen dissolution into the bloodstream, surpassing levels achievable at sea level. The pressure will be raised incrementally, followed by HBOT sessions lasting for a total of 90 minutes. The 90-minute sessions include brief 5-minute intervals for ambient air every 20 minutes to ensure safety and comfort. Treatment will be conducted five days a week over eight weeks.
  Supervised by competent healthcare professionals, HBOT is considered safe, with potential side effects primarily stemming from heightened pressure and, in rare cases, oxygen toxicity.

SUMMARY:
The objective of this observational study is to document symptom progression in 60 patients with myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) who undergo Hyperbaric Oxygen Therapy (HBOT) following COVID or other infections. Participants will receive HBOT treatment as an additional option after completing the Chronic Fatigue Syndrome CARE (CFS_CARE) study and will be invited to take part in this observational study. Patients will complete health evaluations in the form of questionnaires, including the 36-Item Short Form Health Survey (SF-36), to assess changes in ME/CFS-related symptoms after HBOT. Rather than evaluating the efficacy of HBOT itself, the study will focus on observing and documenting these changes. Its goal is to offer valuable insights into symptom progression in ME/CFS patients receiving HBOT, which can serve as a foundation for future interventional randomized controlled trials.

DETAILED DESCRIPTION:
Following mild to moderate COVID infection, around 10% of individuals develop post-COVID syndrome (PCS) characterized by symptoms like fatigue, exercise intolerance, cognitive impairment, headaches, and muscle pain (Kedor et al., 2022). Some PCS patients may later be diagnosed with ME/CFS, a severe and chronic disease triggered by infections (Renz-Polster & Scheibenbogen, 2022). ME/CFS presents symptoms such as debilitating fatigue, exercise intolerance, post-exertional malaise (PEM), headaches, muscle pain, cognitive impairment ("brain fog"), orthostatic intolerance, autonomic dysfunction, sleep disturbances, and a general feeling of illness. Currently, no curative therapy for ME/CFS exists. Therapeutic procedures for ME/CFS mainly focus on symptom management, but evidence-based and standardized treatments are urgently needed due to the high number of patients and the impact on healthcare (Renz-Polster & Scheibenbogen, 2022). Off-label drug and non-drug approaches are used, but their effectiveness lacks sufficient evidence from controlled trials.

ME/CFS and PCS may have different underlying pathomechanisms, with some patients showing endothelial dysfunction and reduced blood flow (Haffke et al., 2022). Enhancing blood flow and promoting the formation of new capillaries is a potential therapeutic approach due to the presumed role of reduced blood flow. In this regard, Hyperbaric Oxygen Therapy (HBOT) is under investigation as a treatment for ME/CFS and PCS, showing promising results in trials (e.g., Zilberman-Itskovich et al., 2022; Robbins et al., 2021; Kjiellberg et al., 2022; Akarsu et al., 2013). This non-interventional observational study aims to document symptom progression in 60 patients with ME/CFS who underwent HBOT following COVID or other infections. The study does not focus on evaluating the efficacy of HBOT itself.

ME/CFS patients currently participating in the Chronic Fatigue Syndrome CARE (CFS_CARE) study at Klinik Bavaria in Kreischa will have the opportunity to receive HBOT treatment as a supplementary offer from the clinic upon completion of the CFS_CARE study. Additionally, these patients will be invited to participate in this observational study during the final CFS_CARE presentation at the 12-month mark. HBOT is performed as part of the Conformité Européenne (CE) certificate, as an outpatient procedure within standard clinical practice, and independent of the study focus. Throughout the HBOT treatment, patients will undergo health assessments and symptom evaluations four weeks after treatment initiation and four weeks after completing the HBOT sessions. To facilitate this, patients will receive a link to a RedCap file containing questionnaires, including those previously utilized in the CFS_CARE study (36-Item Short Form Health Survey (SF-36), Munich Berlin Symptom Questionnaire (MBSQ), Chalder Fatigue Questionnaire, Bell Score). Completing the questionnaires typically requires approximately 45 minutes. The questionnaires will be collected every two months over 12 months, resulting in a total follow-up period of 10 months. A follow-up visit at the outpatient clinic is scheduled for four weeks after HBOT is completed.

The study's primary endpoint is to identify improvements in physical function following HBOT. This will be achieved by utilizing the SF-36 Physical Function (PF) questionnaire, which commonly serves as the primary endpoint in clinical trials focused on ME/CFS. It has been shown that an increase of at least 10 points in the SF-36 PF (range 0 - 100 = healthy) defines clinically relevant improvement ("a little better"), and an increase of 20 points defines greater clinical improvement ("much better") (Brigden 2018). Therefore, an increase of at least 10 points 4 weeks after HBOT is defined as a response and assessed as the primary endpoint.

The study-related measures do not pose significant risks or additional burdens to participants aside from the time required to complete the questionnaires. However, it has the potential to generate valuable knowledge regarding HBOT as a potential treatment for ME/CFS. To date, there has been no documentation of the efficacy of HBOT in ME/CFS through a clinical trial employing objective methods. The results of this observational study are expected to serve as the foundation for a potential interventional randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 18 and 65 years who have previously participated in the CFS_CARE study and have been diagnosed with ME/CFS
* ME/CFS diagnosis based on the Canadian Consensus Criteria (CCC), characterized by exercise intolerance and symptom worsening lasting for a minimum of 14 hours
* Disease severity determined by a Bell Score ranging from 30 to 70
* Plan to undergo 20 or 40 days of Hyperbaric Oxygen Therapy (HBOT)
* Consent provided by the patient

Exclusion Criteria:

* Unwillingness to consent to the storage of pseudonymized clinical data as a part of the study
* Pregnancy
* Presence of medical conditions that could potentially pose a risk during Hyperbaric Oxygen Therapy (HBOT) (e.g., heart failure, pulmonary disease, major depression, panic attacks)
* Acute infection (e.g., COVID, HIV, or hepatitis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty male or female patients, aged between 18 and 65 years, will be included in the study. ME/CFS patients currently participating in the CFS_CARE study through the Bavaria Clinic in Kreischa will have the opportunity to receive HBOT treatment as an additional option provided by the clinic upon completion of the CFS_CARE study. Additionally, these patients will be invited to participate in this observational study during the final CFS_CARE presentation at the 12-month mark.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Physical Function (PF) as measured by the Short Form 36 Health Survey Questionnaire (SF-36). | 4 weeks after completion of HBOT therapy
  The Short Form 36 Health Survey (SF-36) is an established and widely used health-related quality of life measure. The Physical Function (PF) domain asks patients to report limitations on ten mobility activities, such as walking specified distances, carrying groceries, and bathing or dressing. Scores are weighted and transformed into a scale ranging from 0 (greatest possible health restrictions, i.e., severe disability) to 100 (no health restrictions). An intra-patient change of 10 points in SF-36-PF from baseline to week four is considered clinically meaningful.

SECONDARY OUTCOMES:
Duration of improvement in Physical Function (PF) as measured by the Short Form 36 Health Survey Questionnaire (SF-36) | Collected every 2 months over a total of 12 months after completion of HBOT therapy
  Duration of the effect of HBOT therapy as assessed by SF-36 PF. Intra-patient change in physical and mental fatigue from baseline to follow-up points will be documented as indexed by the SF-36 PF.
Improvement in physical and mental fatigue as measured by the Chalder Fatigue Scale | Collected every 2 months over a total of 12 months after completion of HBOT therapy
  The Chalder Fatigue Scale measures the extent and severity of tiredness and has been used in multiple randomized trials of behavioral interventions in patients with ME/CFS. Each of the 11 items is answered on a 4-point scale with an overall score ranging from 0 (asymptomatic) to 33 (maximum symptomology). Intra-patient change in physical and mental fatigue from baseline to follow-up points will be documented as indexed by the Chalder Fatigue Scale.
Improvement in functional disability as measured by the Bell disability scale | Collected every 2 months over a total of 12 months after completion of HBOT therapy
  The Bell disability scale is a standard assessment in ME/CFS that evaluates functional ability in adult ME/CFS patients. Eleven statements describe patient status such as level of symptoms at rest, level of symptoms with exercise, activity level, and ability to perform work, travel and self care. Its score ranges from 0 (bedridden) to 100 (no symptoms). Intra-patient change from baseline to follow-up points will be documented as indexed by the Bell score.
Improvement in disease severity based on self- reported symptoms as measured by the Munich Berlin Symptom Questionnaire (MBSQ) | Collected every 2 months over a total of 12 months after completion of HBOT therapy
  The Munich Berlin Symptom Questionnaire (MBSQ) is a questionnaire for ME/CFS that captures the Institute of Medicine (IOM) and Canadian Consensus Criteria (CCC) as well as a total of 44 symptoms from 8 domains on a scale of 0 - 4 for frequency and severity. From this, a score for total symptom severity ranging from 0 (not present) to 352 (very severe) is calculated. Intra-patient change from baseline to follow-up points will be documented as indexed by the MBSQ.
Improvement in muscle strength as measured by the hand grip strength (HGS) test | 4 weeks after completion of HBOT therapy
  The Hand Grip Strength (HGS) test is a simple yet effective measurement of muscular strength. It involves gripping a dynamometer (or other grip strength measurement device) with maximal force using the dominant hand. The device measures exerted force in kilograms or pounds. Hand grip strength reflects overall muscle strength providing insights into a person's physical health, functional capacity, and potential muscular deficiencies. Intra-patient change in hand grip strength (HGS) from baseline to week four.
Assessment and documentation of tolerability | On the day of completion of HBOT therapy
  Assessment and documentation of tolerability with a questionnaire that is collected at the end of the HBOT therapy
Improvement in orthostatic tolerance as measured by the National Aeronautics and Space Administration (NASA) 10 Minute Lean Test | 4 weeks after completion of HBOT therapy
  The NASA 10-Minute Lean Test evaluates a person's susceptibility to gravitational effects. In post-COVID ME/CFS research, it probes cardiovascular and autonomic nervous system issues stemming from a SARS-CoV-2 infection. During the test, an person lies flat on their back with a slightly elevated head, while blood pressure and heart rate are monitored during a controlled tilt to a head-down position. In about 10 minutes, this provides valuable insights into cardiovascular adaptability and potential dysregulation, aiding understanding of symptoms like dizziness, fatigue, and palpitations in long-COVID patients. Intra-patient change in the NASA 10 Minute Lean Test from baseline to week four.
Improvement in exercise capacity measured by the 1-Minute Sit-to-Stand Test | 4 weeks after completion of HBOT therapy
  The 1-Minute Sit-to-Stand Test is a validated and reliable test for quantifying exercise capacity. In this test, the person starts in a seated position and is instructed to stand up and sit down as many times as possible within a one-minute period. The test provides valuable insights into a person's muscle strength, endurance, and overall physical fitness. Intra-patient change in the 1-minute Sit-to-Stand Test from baseline to week four.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Scheibenbogen, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kedor C, Freitag H, Meyer-Arndt L, Wittke K, Hanitsch LG, Zoller T, Steinbeis F, Haffke M, Rudolf G, Heidecker B, Bobbert T, Spranger J, Volk HD, Skurk C, Konietschke F, Paul F, Behrends U, Bellmann-Strobl J, Scheibenbogen C. A prospective observational study of post-COVID-19 chronic fatigue syndrome following the first pandemic wave in Germany and biomarkers associated with symptom severity. Nat Commun. 2022 Aug 30;13(1):5104. doi: 10.1038/s41467-022-32507-6. PMID 36042189
- [Background] Renz-Polster H, Scheibenbogen C. [Post-COVID syndrome with fatigue and exercise intolerance: myalgic encephalomyelitis/chronic fatigue syndrome]. Inn Med (Heidelb). 2022 Aug;63(8):830-839. doi: 10.1007/s00108-022-01369-x. Epub 2022 Jul 13. German. PMID 35925074
- [Background] Haffke M, Freitag H, Rudolf G, Seifert M, Doehner W, Scherbakov N, Hanitsch L, Wittke K, Bauer S, Konietschke F, Paul F, Bellmann-Strobl J, Kedor C, Scheibenbogen C, Sotzny F. Endothelial dysfunction and altered endothelial biomarkers in patients with post-COVID-19 syndrome and chronic fatigue syndrome (ME/CFS). J Transl Med. 2022 Mar 22;20(1):138. doi: 10.1186/s12967-022-03346-2. PMID 35317812
- [Background] Zilberman-Itskovich S, Catalogna M, Sasson E, Elman-Shina K, Hadanny A, Lang E, Finci S, Polak N, Fishlev G, Korin C, Shorer R, Parag Y, Sova M, Efrati S. Hyperbaric oxygen therapy improves neurocognitive functions and symptoms of post-COVID condition: randomized controlled trial. Sci Rep. 2022 Jul 12;12(1):11252. doi: 10.1038/s41598-022-15565-0. PMID 35821512
- [Background] Robbins T, Gonevski M, Clark C, Baitule S, Sharma K, Magar A, Patel K, Sankar S, Kyrou I, Ali A, Randeva HS. Hyperbaric oxygen therapy for the treatment of long COVID: early evaluation of a highly promising intervention. Clin Med (Lond). 2021 Nov;21(6):e629-e632. doi: 10.7861/clinmed.2021-0462. PMID 34862223
- [Background] Kjellberg A, Abdel-Halim L, Hassler A, El Gharbi S, Al-Ezerjawi S, Bostrom E, Sundberg CJ, Pernow J, Medson K, Kowalski JH, Rodriguez-Wallberg KA, Zheng X, Catrina S, Runold M, Stahlberg M, Bruchfeld J, Nygren-Bonnier M, Lindholm P. Hyperbaric oxygen for treatment of long COVID-19 syndrome (HOT-LoCO): protocol for a randomised, placebo-controlled, double-blind, phase II clinical trial. BMJ Open. 2022 Nov 2;12(11):e061870. doi: 10.1136/bmjopen-2022-061870. PMID 36323462
- [Background] Akarsu S, Tekin L, Ay H, Carli AB, Tok F, Simsek K, Kiralp MZ. The efficacy of hyperbaric oxygen therapy in the management of chronic fatigue syndrome. Undersea Hyperb Med. 2013 Mar-Apr;40(2):197-200. PMID 23682549